CLINICAL TRIAL: NCT05790681
Title: A Study Investigating the Pharmacokinetic Properties of Insulin Icodec in Children and Adolescents With Type 2 Diabetes
Brief Title: A Study to Test How New Long-acting Insulin (Insulin Icodec) Works in the Body of Children and Teenagers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4888; U1111-1271-9231 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Type 2 Diabetes (Experimental): Participants will receive single subcutaneous (s.c.) fixed dose of insulin icodec (700 units per milliliter [U/mL]) that is 5.6 units per kilogram (U/kg) bodyweight. Subjects will be followed up for 5 weeks after dosing.
  Interventions: Drug: Insulin icodec

INTERVENTIONS:
Drug: Insulin icodec — Participants will receive subcutaneously fixed dose of insulin icodec (700 U/mL) that is 5.6 U/kg bodyweight.

SUMMARY:
Insulin icodec is a new medicine which is under development for use in humans and is not yet available at the pharmacy. It is being developed for the treatment of diabetes, a condition that causes high blood sugar levels. Insulin icodec will be investigated in participants with type 2 diabetes. Participant will get one dose of insulin icodec, which will be administered in the afternoon or evening of the day of dosing. The study will last for about 8 weeks. Insulin icodec will be injected into a skin fold with a small needle (subcutaneous application) using a pen injector prefilled with a volume of 3 milliliter (mL) (a little less than a quarter of a teaspoonful). The amount of insulin icodec participant will receive depends on participant's body weight. Participant must not participate if participant meets certain conditions called exclusion criteria, such as an age of above 18 years when the informed consent is signed or has serious health conditions. Female participant cannot take part if she is pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 10 to less than (<) 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus greater than or equal to (>=) 30 days prior to the day of screening
* Glycated haemoglobin (HbA1c) less than or equal to (<=) 10% (86 millimoles per mole [mmol/mol]) at screening
* Treated with basal insulin, premix insulin or continuous subcutaneous insulin infusion (CSII) with or without bolus insulin or additional anti-diabetic drug(s).
* Current daily basal insulin treatment >= 0.2 (I) units per kilogram per day (U/kg/day) with stable doses >=30 days prior to the day of screening

Exclusion Criteria:

* Known or suspected hypersensitivity to study interventions or related products
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin icodec concentration-time curve after a single dose (AUCIco,0-inf,SD) | From 0 hours until infinity after trial product administration (day 1)
  Measured in picomoles*hours per liter (pmol*h/L).
Maximum observed serum insulin icodec concentration after a single dose (Cmax,Ico,SD) | From 0 hours until last measurement time after trial product administration (day 1)
  Measured in picomoles per liter (pmol/L).
Time to maximum observed serum insulin icodec concentration after a single dose (tmax,Ico,SD) | From 0 hours until last measurement time after trial product administration (day 1)
  Measured in hours.

SECONDARY OUTCOMES:
Model-based maximum serum insulin icodec concentration during one dosing interval at steady state (Cmax,Ico,SS,model) | From 0 to 168 hours after trial product administration
  Measured in pmol/L.
Model-based area under the serum insulin icodec concentration-time curve during one dosing interval at steady state (AUC,Ico,τ,SS,model) | From 0 to 168 hours after trial product administration
  Measured in pmol*h/L.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (13):
- United States (13):
  - Children's Hosp-Los Angeles, Los Angeles, California
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Yale New Haven Hospital, Hospital Research Unit, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Nemours Children's Health, Jacksonville, Florida
  - Nemours Chld Clnc Jacksonville, Jacksonville, Florida
  - Pennington Biom Res Ctr, Baton Rouge, Louisiana
  - John Hopkins Univ Hosp, Baltimore, Maryland
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - Cincinnati Child's Hsp Med Ctr, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Virginia Clinical Research Unit, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on NovoNordisk-trials.com
URL: http://novonordisk-trials.com